CLINICAL TRIAL: NCT02246504
Title: Registry - Use of a High Intensity Focused Ultrasound (HIFU) in Patients With Non-malignant Thyroid Nodules.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theraclion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFU/BG/NT
Record Dates: First submitted 2014-09-16; First posted 2014-09-22 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Non-malignant Thyroid Nodule

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HIFU treatment (Experimental): use of HIFU treatment in patients with non-malignant thyroid nodules
  Interventions: Device: HIFU treatment

INTERVENTIONS:
Device: HIFU treatment

SUMMARY:
The purpose of this study is to evaluate thyroid nodule's volume, structure and vascularisation changes following HIFU therapy assessed by ultrasonography

DETAILED DESCRIPTION:
HIFU treatment will be performed under conscious sedation under the supervision / responsibilities of an anesthetist.

A maximum of 2 HIFU sessions per nodule will be performed per patient. The decision to retreat the patient will be taken at 1 month post-HIFU or later.

Follow-up after HIFU treatment

D1 after HIFU session:

* Indirect laryngoscopy to check vocal cord mobility.

D7 after HIFU session

* Clinical examination (skin, local symptoms, oedema, voice….),
* Ultrasonography and Power Doppler,

M1 after HIFU session

* Clinical examination (skin, local symptoms, oedema, voice….),
* Ultrasonography and Power Doppler,

M3 after HIFU session

* Clinical examination (skin, local symptoms, oedema, voice….),
* Ultrasonography and Power Doppler Decision for an additional HIFU course to improve volume reduction.

In case of a second HIFU session D7b, M1b and M3b, M6b, M9b, M12b, M18b, M24b and M36b will be performed

M6 after last HIFU session

* Clinical examination (skin, local symptoms, oedema, voice….),
* Ultrasonography and Power Doppler
* TSH
* Free T4
* Antithyroid peroxidase antibodies
* Calcemia and PTH (in case of bilateral treatment or in case previous thyroid surgery)

M9 after HIFU session

* Clinical examination (skin, local symptoms, oedema, voice….),
* Ultrasonography and Power Doppler

M12 after last HIFU session

* Clinical examination (skin, local symptoms, oedema, voice….),
* Ultrasonography and Power Doppler
* TSH
* Free T4
* Antithyroid peroxidase antibodies
* Calcemia and PTH (in case of bilateral treatment or in case previous thyroid surgery)

M18, M24, M36 after HIFU session

* Clinical examination (skin, local symptoms, oedema, voice….),
* Ultrasonography and Power Doppler

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient 18 years or older.
* Patient presenting with at least one thyroid nodule with no signs of malignancy:

  1. Non suspect clinically and at ultrasonography imaging
  2. Benign cytological diagnosis at FNAB from the last 6 months
  3. Normal serum calcitonin
  4. No history of neck irradiation
* Normal TSH.
* Targeted nodule accessible and eligible to HIFU
* Absence of abnormal vocal cord mobility at laryngoscopy.
* Nodule diameter ≥ 10mm measured by ultrasound.
* Composition of the targeted nodule(s) : no more than 30% cystic

Exclusion Criteria:

* Head and/or neck disease that prevents hyperextension of neck.
* Known history of thyroid cancer or other neoplasias in the neck region.
* History of neck irradiation.
* Macrocalcification inducing a shadow in the thyroid significant enough to preclude the HIFU treatment
* Posterior position of the nodule if the thickness of the nodule is <15mm
* Pregnant or lactating woman
* Any contraindication to IV neurolept analgesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10-09 (Actual); Primary Completion 2017-03-07 (Actual); Study Completion 2017-03-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in thyroid nodule's volume | Month 6

SECONDARY OUTCOMES:
Change from baseline in thyroid nodule's structure and vascularisation | Month 6
Number of participants with adverse events | D1, D7, M1, M3 and M6

CONTACTS AND LOCATIONS:
Overall Officials: Roussanka Kovatcheva, Prof., Principal Investigator
Locations (1):
- Clinic of thyroid and metabolite bone disease of the Acad. of Ivan Penchev UDHATE - 2, Zdrave street, Sofia, Bulgaria